CLINICAL TRIAL: NCT05010707
Title: Effectiveness and Safety of Different Estradiol Replacement Therapies in Transgender Female
Brief Title: Transgender Estradiol Affirming Therapy
Acronym: TREAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ginger E Nicol, Associate Professor of Child & Adolescent Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202104092
Record Dates: First submitted 2021-07-16; First posted 2021-08-18 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Transgenderism
Keywords: Transgender female; Gender affirming hormone therapy; Estrogen therapy
MeSH Terms: conditions — Transsexualism | interventions — Transdermal Patch; Spironolactone

STUDY DESIGN:
Intervention Model Description: Participants who agreed to be in the study will undergo block randomization into three groups:
  1. daily sublingual 17 beta estradiol
  2. twice daily sublingual 17 beta estradiol
  3. transdermal 17 beta estradiol
  All patients will also receive spironolactone as antiandrogen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transdermal estradiol plus spironolactone (Active Comparator): Starting dose will be 100 mcg/24hrs Plan to increase by 100 mcg/24hrs every month to a max dose of 400 mcg/24hrs Goal is to achieve a serum estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels
  All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Interventions: Drug: Transdermal patch; Diagnostic Test: Pro-thrombotic markers; Diagnostic Test: Metabolic markers; Diagnostic Test: Hormone Profile; Drug: Spironolactone
- Daily sublingual estradiol plus spironolactone (Active Comparator): Starting dose will be 2 mg daily Plan to increase every month by 2 mg daily Goal is to achieve serum estradiol level between 100-200 pg/mL mL and to suppress testosterone to cisgender female levels.
  All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Interventions: Diagnostic Test: Pro-thrombotic markers; Diagnostic Test: Metabolic markers; Diagnostic Test: Hormone Profile; Drug: Daily Sublingual Tablet; Drug: Spironolactone
- Twice daily sublingual estradiol plus spironolactone (Active Comparator): Starting dose will be 1 mg twice daily Plan to increase every month by 2 mg daily divided BID Goal is to achieve serum estradiol level between 100-200 pg/mL mL and to suppress testosterone to cisgender female levels
  All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Interventions: Diagnostic Test: Pro-thrombotic markers; Diagnostic Test: Metabolic markers; Diagnostic Test: Hormone Profile; Drug: BID Sublingual Tablet; Drug: Spironolactone

INTERVENTIONS:
Drug: Transdermal patch — Participants will be prescribed the medication and dosed based on their hormonal profile. Goal is achieve estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels
  Other Names: Daily
  Arms: Transdermal estradiol plus spironolactone
Diagnostic Test: Pro-thrombotic markers — Once participants are started on gender affirming hormone therapy, pro-thombotic markers will be checked at baseline and every 6 months. Pro-thrombotic markers will include: Factor II, Factor IX, Factor XI, Von Willebrand factor, Protein C, Protein S, activated Protein C resistance.
Diagnostic Test: Metabolic markers — Once participants are started on gender affirming hormone therapy, metabolic markers will be checked at baseline and every 6 months. Markers will include: Insulin level, fasting glucose, body mass index, waist circumference.
Diagnostic Test: Hormone Profile — Once participants are started on gender affirming hormone therapy, hormonal levels will be checked every 4 weeks until estradiol and testosterone levels are within goal as established by standard of care.
Drug: Daily Sublingual Tablet — Participants will be prescribed the medication and dosed based on their hormonal profile. Participants will take dose as once daily medication. Goal is achieve estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels
  Other Names: Once daily dosing
  Arms: Daily sublingual estradiol plus spironolactone
Drug: BID Sublingual Tablet — Participants will be prescribed the medication and dosed based on their hormonal profile. Participants will take dose as twice daily medication. Goal is achieve estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels
  Other Names: Twice daily dosing
  Arms: Twice daily sublingual estradiol plus spironolactone
Drug: Spironolactone — All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Other Names: Daily

SUMMARY:
The purpose of this open label, pilot, randomized clinical trial is to evaluate the effectiveness, safety and tolerability of estrogen use in transgender female and the degree of testosterone suppression achieved in this population when placed on gender affirming pharmacological therapy.

DETAILED DESCRIPTION:
Transgender patients suffer from poor mental and medical health outcomes compared to their cisgender peers. Given the widespread acknowledgment of the health care needs of transgender people, priority should be given to those actions that will ensure safe and appropriate care in health centers.

The current hormone therapy is not uniform and depends on the health care system, cost considerations, and differences in the regional availability of estrogens and antiandrogens. A typical regimen includes estrogen to provide feminizing effects in conjunction with therapy to block testosterone (antiandrogens or gonadotropin-releasing hormone [GnRH] analogs). Estrogen also inhibits testosterone secretion.

Ethinyl estradiol was previously the mainstay of most estrogen-directed therapies; this is no longer the case due to its increased risk of cardiovascular death and increased incidence of deep venous thrombosis. 17-beta estradiol, which can be provided in tablet, patch, and injection, is currently the preferred formulation.

This open label, pilot, randomized clinical trial will evaluate the effectiveness and safety of gender affirming hormone therapy with estrogen and the degree of testosterone suppression achieved in transgender female patients when placed on daily sublingual 17-beta estradiol, twice daily sublingual 17-beta estradiol, or transdermal 17-beta estradiol. All patients will also receive spironolactone as antiandrogen.

One of the major complications from estradiol GAHT is thromboembolism. The investigators will also determine the effects of the different estradiol regimens on thrombosis markers. These studies will be the first to determine if the dosing regimen of estradiol affects risk markers in transgender women.

ELIGIBILITY:
Inclusion Criteria:

* Female transgender patients between the ages of 18 to 30 years of age who are seen at the Washington University Transgender Center. Patients must have met the eligibility and readiness criteria for gender-affirming hormone therapy.

Exclusion Criteria:

* GnRH agonist for the last 12 months
* History of liver disease
* Dyslipidemia requiring treatment
* Cigarette smoking
* Body mass index >30 kg/m2

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female gender identity
Enrollment: 39 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginger Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Transgender Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Unger CA. Hormone therapy for transgender patients. Transl Androl Urol. 2016 Dec;5(6):877-884. doi: 10.21037/tau.2016.09.04. PMID 28078219
- [Background] Kaltiala-Heino R, Bergman H, Tyolajarvi M, Frisen L. Gender dysphoria in adolescence: current perspectives. Adolesc Health Med Ther. 2018 Mar 2;9:31-41. doi: 10.2147/AHMT.S135432. eCollection 2018. PMID 29535563
- [Background] Connolly MD, Zervos MJ, Barone CJ 2nd, Johnson CC, Joseph CL. The Mental Health of Transgender Youth: Advances in Understanding. J Adolesc Health. 2016 Nov;59(5):489-495. doi: 10.1016/j.jadohealth.2016.06.012. Epub 2016 Aug 17. PMID 27544457
- [Background] Hamidi O, Davidge-Pitts CJ. Transfeminine Hormone Therapy. Endocrinol Metab Clin North Am. 2019 Jun;48(2):341-355. doi: 10.1016/j.ecl.2019.02.001. Epub 2019 Mar 23. PMID 31027544
- [Background] Asscheman H, Giltay EJ, Megens JA, de Ronde WP, van Trotsenburg MA, Gooren LJ. A long-term follow-up study of mortality in transsexuals receiving treatment with cross-sex hormones. Eur J Endocrinol. 2011 Apr;164(4):635-42. doi: 10.1530/EJE-10-1038. Epub 2011 Jan 25. PMID 21266549
- [Background] Angus LM, Nolan BJ, Zajac JD, Cheung AS. A systematic review of antiandrogens and feminization in transgender women. Clin Endocrinol (Oxf). 2021 May;94(5):743-752. doi: 10.1111/cen.14329. Epub 2020 Oct 5. PMID 32926454
- [Background] Spanos C, Bretherton I, Zajac JD, Cheung AS. Effects of gender-affirming hormone therapy on insulin resistance and body composition in transgender individuals: A systematic review. World J Diabetes. 2020 Mar 15;11(3):66-77. doi: 10.4239/wjd.v11.i3.66. PMID 32180895
- [Background] Bagot CN, Marsh MS, Whitehead M, Sherwood R, Roberts L, Patel RK, Arya R. The effect of estrone on thrombin generation may explain the different thrombotic risk between oral and transdermal hormone replacement therapy. J Thromb Haemost. 2010 Aug;8(8):1736-44. doi: 10.1111/j.1538-7836.2010.03953.x. Epub 2010 Jun 14. PMID 20553380
- [Background] Hembree WC, Cohen-Kettenis PT, Gooren L, Hannema SE, Meyer WJ, Murad MH, Rosenthal SM, Safer JD, Tangpricha V, T'Sjoen GG. Endocrine Treatment of Gender-Dysphoric/Gender-Incongruent Persons: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2017 Nov 1;102(11):3869-3903. doi: 10.1210/jc.2017-01658. PMID 28945902
- [Background] Bao AM, Liu RY, van Someren EJ, Hofman MA, Cao YX, Zhou JN. Diurnal rhythm of free estradiol during the menstrual cycle. Eur J Endocrinol. 2003 Feb;148(2):227-32. doi: 10.1530/eje.0.1480227. PMID 12590642
- [Derived] Cortez S, Moog D, Lewis C, Williams K, Herrick C, Fields M, Gray T, Guo Z, Nicol G, Baranski T. Effectiveness and Safety of Different Estradiol Regimens in Transgender Women (TREAT Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 22;12:e53092. doi: 10.2196/53092. PMID 38133914

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Estradiol Plus Spironolactone: Starting dose will be 100 mcg/24hrs Plan to increase by 100 mcg/24hrs every month to a max dose of 400 mcg/24hrs Goal is to achieve a serum estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels
  All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Transdermal patch: Participants will be prescribed the medication and dosed based on their hormonal profile. Goal is achieve estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels
  Pro-thrombotic markers: Once participants are started on gender affirming hormone therapy, pro-thombotic markers will be checked at baseline and every 6 months. Pro-thrombotic markers will include: Factor II, Factor IX, Factor XI, Von Willebrand factor, Protein C, Protein S, activated Protein C resistance.
  Metabolic markers: Once participants are started on gender affirming hormone therapy, metabolic markers will be checked at baseline and every 6 months. Markers will include: Insulin level, fasting glucose, body mass index, waist circumference.
  Hormone Profile: Once participants are started on gender affirming hormone therapy, hormonal levels will be checked every 4 weeks until estradiol and testosterone levels are within goal as established by standard of care.
- Daily Sublingual Estradiol Plus Spironolactone: Starting dose will be 2 mg daily Plan to increase every month by 2 mg daily Goal is to achieve serum estradiol level between 100-200 pg/mL mL and to suppress testosterone to cisgender female levels.
  All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Pro-thrombotic markers: Once participants are started on gender affirming hormone therapy, pro-thombotic markers will be checked at baseline and every 6 months. Pro-thrombotic markers will include: Factor II, Factor IX, Factor XI, Von Willebrand factor, Protein C, Protein S, activated Protein C resistance.
  Metabolic markers: Once participants are started on gender affirming hormone therapy, metabolic markers will be checked at baseline and every 6 months. Markers will include: Insulin level, fasting glucose, body mass index, waist circumference.
  Hormone Profile: Once participants are started on gender affirming hormone therapy, hormonal levels will be checked every 4 weeks until estradiol and testosterone levels are within goal as established by standard of care.
  Daily Sublingual Tablet: Participants will be prescribed the medication and dosed based on their hormonal profile. Participants will take dose as once daily medication. Goal is achieve estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels.
- Twice Daily Sublingual Estradiol Plus Spironolactone: Starting dose will be 1 mg twice daily Plan to increase every month by 2 mg daily divided BID Goal is to achieve serum estradiol level between 100-200 pg/mL mL and to suppress testosterone to cisgender female levels
  All patients will also receive spironolactone. Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Spironolactone will be started at 50 mg daily and will increase to standard dose.
  Pro-thrombotic markers: Once participants are started on gender affirming hormone therapy, pro-thombotic markers will be checked at baseline and every 6 months. Pro-thrombotic markers will include: Factor II, Factor IX, Factor XI, Von Willebrand factor, Protein C, Protein S, activated Protein C resistance.
  Metabolic markers: Once participants are started on gender affirming hormone therapy, metabolic markers will be checked at baseline and every 6 months. Markers will include: Insulin level, fasting glucose, body mass index, waist circumference.
  Hormone Profile: Once participants are started on gender affirming hormone therapy, hormonal levels will be checked every 4 weeks until estradiol and testosterone levels are within goal as established by standard of care.
  BID Sublingual Tablet: Participants will be prescribed the medication and dosed based on their hormonal profile. Participants will take dose as twice daily medication. Goal is achieve estradiol level between 100-200 pg/mL and to suppress testosterone to cisgender female levels.
Period: Overall Study
Arm/Group | Transdermal Estradiol Plus Spironolactone | Daily Sublingual Estradiol Plus Spironolactone | Twice Daily Sublingual Estradiol Plus Spironolactone
Started | 12 | 13 | 14
Completed | 11 | 12 | 14
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total number of 39 participants had the demographic information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Estradiol Plus Spironolactone | Daily Sublingual Estradiol Plus Spironolactone | Twice Daily Sublingual Estradiol Plus Spironolactone | Total
Number analyzed (Participants) | 12 | 13 | 14 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 14 | 39
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 25.3 [18.2 to 42.6] | 25.0 [19.0 to 37.2] | 21.5 [18.9 to 33.5] | 25.3 [18.2 to 42.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 14 | 39
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 9 | 12 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 14 | 39
Weight [Mean (Standard Deviation); unit: Kg] | 75.6 (17.2) | 82.1 (20.9) | 74.0 (13.0) | 77.3 (17.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (5.9) | 26.2 (7.2) | 23.9 (5.0) | 25.1 (6.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 132.8 (12.6) | 140.8 (21.7) | 128.3 (16.9) | 134.0 (18.0)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 87.9 (6.7) | 87.5 (9.7) | 82.1 (10.4) | 86.0 (9.0)
Height [Mean (Standard Deviation); unit: cm] | 173.5 (6.5) | 177.6 (9.9) | 176.9 (8.4) | 175.9 (8.4)
Waist circumference [Mean (Standard Deviation); unit: inch] | 34.8 (7.0) | 36 (7.2) | 33.9 (5.2) | 34.9 (6.3)
Lifestyle [Number; unit: participants]
  Alcohol use | 1 | 3 | 1 | 5
  Vaping | 0 | 0 | 2 | 2
Estradiol [Mean (Standard Deviation); unit: pg/mL] | 27.1 (15.5) | 25.8 (10.8) | 23.4 (13.5) | 25.3 (13.0)
Estrone [Mean (Standard Deviation); unit: pg/mL] | 37.2 (20.7) | 27.7 (20.9) | 26.7 (14.0) | 30.2 (18.7)
Total testosterone [Mean (Standard Deviation); unit: ng/dL] | 498.1 (160.6) | 481.3 (230.2) | 505.3 (206.5) | 495.0 (198.1)
Sodium [Mean (Standard Deviation); unit: mmol/L] | 140.3 (2.1) | 140.4 (1.4) | 139.1 (1.6) | 139.9 (1.8)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.0 (0.4) | 4.0 (0.3) | 4.2 (0.5) | 4.1 (0.4)
Chloride [Mean (Standard Deviation); unit: mmol/L] | 103.0 (1.9) | 102.9 (2.4) | 101.6 (2.0) | 102.4 (2.2)
Bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 24.2 (3.1) | 26.0 (2.9) | 25.1 (3.5) | 25.1 (3.2)
Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 14.3 (3.7) | 12.5 (3.2) | 14.1 (5.5) | 13.6 (4.3)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.0 (0.2) | 0.9 (0.1) | 0.9 (0.2) | 0.9 (0.2)
Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.7 (0.3) | 9.6 (0.3) | 9.8 (0.3) | 9.7 (0.3)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.5 (0.3) | 0.5 (0.2) | 0.5 (0.3) | 0.5 (0.3)
Plasma protein [Mean (Standard Deviation); unit: g/dL] | 7.8 (0.3) | 7.7 (0.4) | 7.8 (0.7) | 7.7 (0.5)
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.9 (0.3) | 4.9 (0.3) | 4.9 (0.3) | 4.9 (0.3)
Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] | 82.3 (22.1) | 75.9 (24.0) | 77.6 (17.0) | 78.4 (20.6)
AST [Mean (Standard Deviation); unit: U/L] | 25.2 (6.0) | 23.0 (6.4) | 22.2 (6.6) | 23.3 (6.3)
ALT [Mean (Standard Deviation); unit: U/L] | 30.3 (16.2) | 23.2 (9.7) | 24.1 (14.8) | 25.6 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Testosterone Level in Transgender Female Patients
Description: Degree of testosterone suppression by measuring total testosterone level in transgender female patients undergoing hormonal affirming therapy, clinical testosterone level in pg/mL
Time Frame: Change from baseline total testosterone level at 1 and 6 months
Population: Baseline Measures
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Transdermal Estradiol Plus Spironolactone | Daily Sublingual Estradiol Plus Spironolactone | Twice Daily Sublingual Estradiol Plus Spironolactone
Number analyzed (Participants) | 11 | 13 | 14
pg/mL
  Baseline | 498.6 (46.2) | 481.3 (61.3) | 505.3 (53.2)
  1 Month | 62.7 (13.7) | 278.5 (54.8) | 313.8 (69.7)
  6 Month | 29.4 (7.4) | 108.1 (46.5) | 124.7 (72.5)
Statistical Analysis 1: Comparison: Transdermal Estradiol Plus Spironolactone vs Daily Sublingual Estradiol Plus Spironolactone vs Twice Daily Sublingual Estradiol Plus Spironolactone; Time x treatment (month 0, and 1 month); Test type: Superiority; p = 0.005, Mixed Models Analysis
Statistical Analysis 2: Comparison: Transdermal Estradiol Plus Spironolactone vs Daily Sublingual Estradiol Plus Spironolactone; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = -225.3, 95% CI 2-sided [-421.71 to -28.79]
Statistical Analysis 3: Comparison: Transdermal Estradiol Plus Spironolactone vs Twice Daily Sublingual Estradiol Plus Spironolactone; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = -250.6, 95% CI 2-sided [-447.10 to -54.19]

2. Primary Outcome: Estradiol Level in Transgender Female Patients
Description: Degree of testosterone suppression by measuring estradiol level in transgender female patients affirming hormone therapy
Time Frame: Change from baseline estradiol level at 1 and 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Transdermal Estradiol Plus Spironolactone | Daily Sublingual Estradiol Plus Spironolactone | Twice Daily Sublingual Estradiol Plus Spironolactone
Number analyzed (Participants) | 11 | 13 | 14
pg/mL
  baseline | 28.3 (4.4) | 25.8 (2.9) | 23.4 (3.5)
  1 Month | 56.8 (9.4) | 52.6 (9.6) | 55.2 (5.2)
  6 Months | 74.0 (15.6) | 95.3 (10.5) | 79.4 (11.6)
Statistical Analysis 1: Comparison: Transdermal Estradiol Plus Spironolactone vs Daily Sublingual Estradiol Plus Spironolactone vs Twice Daily Sublingual Estradiol Plus Spironolactone; Time x treatment (month 0 and month 1); Test type: Superiority; p = 0.951, Mixed Models Analysis
Statistical Analysis 2: Comparison: Transdermal Estradiol Plus Spironolactone vs Daily Sublingual Estradiol Plus Spironolactone; Test type: Superiority; p = 1, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-29.6 to 26.4] — The mean difference is computed using the model based estimates rather than from the raw data
Statistical Analysis 3: Comparison: Transdermal Estradiol Plus Spironolactone vs Twice Daily Sublingual Estradiol Plus Spironolactone; Test type: Superiority; p = 1, Mixed Models Analysis; Mean Difference (Final Values) = -7.1, 95% CI 2-sided [-35.1 to 20.8] — The mean difference is computed using the model based estimates rather than from the raw data

3. Primary Outcome: Estrone Level in Transgender Female Patients
Description: Degree of testosterone suppression by measuring estrone level in transgender female patients affirming hormone therapy
Time Frame: Change from baseline estrone level at 1, and 6 months
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Transdermal Estradiol Plus Spironolactone | Daily Sublingual Estradiol Plus Spironolactone | Twice Daily Sublingual Estradiol Plus Spironolactone
Number analyzed (Participants) | 11 | 13 | 14
pg/ml
  baseline | 33.5 (6.8) | 27.7 (5.7) | 26.7 (3.7)
  1 Month | 41.0 (5.2) | 302 (76.1) | 240.1 (36.4)
  6 Months | 57.3 (7.7) | 635.7 (81.3) | 532.9 (124.6)
Statistical Analysis 1: Comparison: Transdermal Estradiol Plus Spironolactone vs Daily Sublingual Estradiol Plus Spironolactone vs Twice Daily Sublingual Estradiol Plus Spironolactone; Time x treatment (month 0 and month 1); Test type: Superiority; p = 0.004, Mixed Models Analysis
Statistical Analysis 2: Comparison: Transdermal Estradiol Plus Spironolactone vs Daily Sublingual Estradiol Plus Spironolactone; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -280.4, 95% CI 2-sided [-487.3 to -73.5]
Statistical Analysis 3: Comparison: Transdermal Estradiol Plus Spironolactone vs Twice Daily Sublingual Estradiol Plus Spironolactone; Test type: Superiority; p = 0.054, Mixed Models Analysis; Mean Difference (Final Values) = -204.1, 95% CI 2-sided [-411.1 to 2.8]

ADVERSE EVENTS:
Time Frame: The time frame is until the study's completion, an average of 12 months.
Arm/Group | Transdermal Estradiol Plus Spironolactone | Daily Sublingual Estradiol Plus Spironolactone | Twice Daily Sublingual Estradiol Plus Spironolactone
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT05010707/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT05010707/ICF_003.pdf